CLINICAL TRIAL: NCT04990648
Title: The Effect of Buzzy® Application on the Pain Level During Vaccine Injection in Infants
Brief Title: Buzzy® Application in Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Ozge Siktas, Principal Investigator, RN, MSc, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-17-02
Record Dates: First submitted 2021-06-30; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Pain; Vaccination; Baby; Buzzy; Pediatric nurse
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buzzy group (Experimental): Buzzy ® was placed on the left arm deltoid muscle site and kept there for 30 seconds. After 30 seconds, Buzzy ® was taken 1 cm up and MMR vaccine injection was administered to the left deltoid muscle site. After the vaccine injection, Buzzy ® was taken to the injection site and kept for another 30 seconds.
  Interventions: Device: Buzzy
- Control group (No Intervention): MMR vaccine injection was administered to the left deltoid muscle without any intervention or application to the injection site.

INTERVENTIONS:
Device: Buzzy — Buzzy ® device (Buzzy ® Mini Healthcare) has been used to reduce pain by using local cold application and vibration effect. Buzzy ® was developed by Dr. Amy Baxter in 2009. The size of the Buzzy ® device measures 2⅞ꞌꞌ x 1⅞ꞌꞌ x ⅞ꞌꞌ (7,2 cm x 4,8 cm x 2,2 cm). It is a bee-shaped device made of hard plastic with a vibrating motor (2 settings - fixed and pulsed), powered by a 2AAA battery. There are 4 ice packages and elastic fastening strap. On the part where the device touches the skin, there is an ice package in the shape of a wing. When the button on the device is pressed, it vibrates.
  Arms: Buzzy group

SUMMARY:
The research was conducted as a randomized controlled experiment to investigate the effect of Buzzy® on pain level during the measles-rubella-mumps (MMR) vaccine injection in 12-month-old infants. This study was done with infants meeting the sampling criteria (buzzy group: 30, control group: 30) on November 2018-May 2019 in Istanbul Bakirkoy 9 Family Health Center.

DETAILED DESCRIPTION:
To determine the effect of Buzzy® application on pain, which is a combination of cold and vibration, during measles-rubella-mumps (MMR) vaccine injection administration on 12-month-old infants. The study is a randomized contrlled experimental research. The research sample is composed of 60 infants (buzzy:30, control:30) who are 12-month-old injected MMR vaccine at Bakırköy No. 9 Family Health Center between November 2018-May 2019. As a data collection tool Data Collection Form, FLACC Pain Scale and Buzzy® device have been used. While Buzzy® was applied on infants in the trial group before, during and after the vaccine injection, the infants in the control group were applied routine vaccine injection. The pain response of the infants was evaluated by the nurse and the parent before, during and after the vaccine injection and the physiological parameters were evaluated by the nurse before and after the vaccine injection.

ELIGIBILITY:
Inclusion Criteria:

* The baby has completed 12 months,
* MMR vaccine will be applied,
* Being at a suitable weight for the month,
* The baby has not been given analgesic medication during the day,
* It can be listed as the parent's willingness to participate in the research.

Exclusion Criteria:

* It can be listed as having a body temperature above 37.5.

Ages: 12 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
The effect of Buzzy® administered during vaccine injection on the infant's pain level before vaccine injection. | 30 seconds
  FLACC Pain Scale was used for determain pain level in this research. Scale got 0 to 10 points (0 (Good) to 10 (Bad)).
The effect of Buzzy® administered during vaccine injection on the infant's pain level during vaccine injection. | 30 seconds
  FLACC Pain Scale was used for determain pain level in this research. Scale got 0 to 10 points (0 (Good) to 10 (Bad)).
The effect of Buzzy® administered during vaccine injection on the infant's pain level after vaccine injection. | 30 seconds
  FLACC Pain Scale was used for determain pain level in this research. Scale got 0 to 10 points (0 (Good) to 10 (Bad)).
The effect of Buzzy® administered during vaccine injection on the infant's pulse before vaccine injection. | 30 seconds
  pulse rate
The effect of Buzzy® administered during vaccine injection on the infant's pulse after vaccine injection. | 30 seconds
  pulse rate
The effect of Buzzy® administered during vaccine injection on infant blood pressure before vaccine injection. | 30 seconds
  blood pressure
The effect of Buzzy® administered during vaccine injection on infant blood pressure after vaccine injection. | 30 seconds
  blood pressure
The effect of Buzzy® administered during vaccine injection on the infant's SpO2 before vaccine injection. | 30 seconds
  SpO2
The effect of Buzzy® administered during vaccine injection on the infant's SpO2 after vaccine injection. | 30 seconds
  SpO2

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University, Tuzla, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No